CLINICAL TRIAL: NCT02716909
Title: Pessary in Singleton Gestations With Short Cervix Without Prior Preterm Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Medical Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 213/2015
Record Dates: First submitted 2016-03-06; First posted 2016-03-23 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical Pessary (Experimental): The cervical pessary is a silicone device that has been used to prevent SPTB Pessary will be placed between 18 and 23 6/7 weeks gestation, and will be removed during the 37th week of pregnancy (or earlier, if indicated)
  Interventions: Device: Cervical pessary
- No intervention (No Intervention): No pessary No pessary will be used. Subjects will receive standard obstetrical management

INTERVENTIONS:
Device: Cervical pessary — The cervical pessary is a silicone device that has been used to prevent SPTB Pessary will be placed between 18 and 23 6/7 weeks gestation, and will be removed during the 37th week of pregnancy (or earlier, if indicated)
  Arms: Cervical Pessary

SUMMARY:
Spontaneous preterm birth (SPTB) remains the number one cause of perinatal mortality in many countries, including the United States. In singleton gestations a short cervical length (CL) on transvaginal ultrasound (TVU) has been shown to be a good predictor of SPTB.

The cervical pessary is a silicone device that has been used to prevent SPTB. The efficacy of cervical pessary has been assessed in several populations including singletons with short CL, unselected twins, twins with a short CL, and triplet pregnancies. Several randomized clinical trials (RCTs) have been published, and several are ongoing. However, no consensus on the use of cervical pessary in pregnancy or guidelines for management have been assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Singleton pregnancy (limits the participants to female gender)
* Short cervical length (less than or equal to 25 mm) on second trimester transvaginal ultrasound at 18-23 6/7 weeks gestation

Exclusion Criteria:

* Multiple gestation
* Prior spontaneous preterm birth 16-36 6/7 weeks
* Ruptured membranes
* Lethal fetal structural anomaly
* Fetal chromosomal abnormality
* Cerclage in place (or planned placement)
* Vaginal bleeding
* Suspicion of chorioamnionitis
* Ballooning of membranes outside the cervix into the vagina or CL = 0 mm on transvaginal ultrasound
* Painful regular uterine contractions
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Spontaneous preterm birth (SPTB) <34 weeks | Less than 34 weeks gestation
  Spontaneous preterm delivery less than 34 weeks of gestation

SECONDARY OUTCOMES:
SPTB <37w | Less than 37 weeks gestation
SPTB <32w | Less than 32 weeks gestation
SPTB <28w | Less than 32 weeks gestation
Gestational age at delivery | Time of delivery
Latency | time of delivery
  interval from randomization to delivery in days
preterm premature rupture of membranes | Less than 34 weeks gestation
Type of delivery | time of delivery
  Cesarean delivery, operative vaginal delivery and spontaneous vaginal delivery
Maternal side effects | Time of delivery
  Vaginal discharge, bacterial vaginosis
Birth weight | Time of delivery
Neonatal death | Between birth and 28 days of age
perinatal death | fetal death after 20 weeks
  either fetal mortality or neonatal death
Composite adverse perinatal outcome | Between birth and 28 days of age
  Includes necrotizing enterocolitis, Intraventricular hemorrhage (grade 3 or higher), respiratory distress syndrome, bronchopulmonary dysplasia (BPD), retinopathy, blood-culture proven sepsis, and neonatal death
Chorioamnionitis | Time of delivery
Adminssion to neonatal intensive care unit | Between birth and 28 days of age

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saccone G, Maruotti GM, Giudicepietro A, Martinelli P; Italian Preterm Birth Prevention (IPP) Working Group. Effect of Cervical Pessary on Spontaneous Preterm Birth in Women With Singleton Pregnancies and Short Cervical Length: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2317-2324. doi: 10.1001/jama.2017.18956. PMID 29260226